CLINICAL TRIAL: NCT05725850
Title: Evaluation of the Effect of an Experimental Gel Based on Jambu Extract ( Acmella Oleracea) in Reducing Post-bleaching Tooth Sensitivity : a Randomized Clinical Study
Brief Title: The Effect of an Experimental Gel Based on Acmella Oleracea Extract in Reducing Post-bleaching Tooth Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Professor of the Graduate Program in Dentistry at the Federal University of Pará, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara-015
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Tooth Bleaching; Pain; Dentin Desensitizing Agents
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EG (Experimental A. Oleracea extract gel) (Experimental): The EG group received the application of experimental gel of A. Oleracea extract for post tooth bleaching sensitivity.
  Interventions: Other: EG (Experimental A. Oleracea extract gel)
- GP (Gel placebo) (Placebo Comparator): The GP group received the application of a placebo gel.
  Interventions: Other: GP (Gel placebo)

INTERVENTIONS:
Other: EG (Experimental A. Oleracea extract gel) — Prior to bleaching treatment with 35% hydrogen peroxide, the dental elements of the EG received application of the experimental desensitizing gel on the buccal surfaces of the central incisors, lateral incisors, canines and upper and lower premolars, with a rubber cup in an active way, for 10 minutes.
  Arms: EG (Experimental A. Oleracea extract gel)
Other: GP (Gel placebo) — Prior to bleaching treatment with 35% hydrogen peroxide, the GP group also received the application of a placebo gel (without active ingredient), under the same conditions described for the experimental gel.
  Arms: GP (Gel placebo)

SUMMARY:
This randomized, double-blind clinical trial aimed to evaluate the effect of an experimental gel containing 10% jambu extract (Acmella Oleracea) in reducing postoperative tooth sensitivity caused by bleaching with 35% hydrogen peroxide. The volunteers of this study were randomized into two different groups - GE (A. Oleracea extract at 10%) and GP (placebo). The dental elements of the GE received application of the experimental desensitizing gel on the buccal surfaces of the central incisors, lateral incisors, canines and upper and lower premolars, with a rubber cup in an active way, for 10 minutes. The GP group also received the application of a placebo gel (without active ingredient), under the same conditions described for the experimental gel. Subsequently, all groups underwent in-office bleaching treatment with 35% hydrogen peroxide.Post-bleaching sensitivity was collected through a form composed of the visual analogue scale (VAS). Color measurement was performed at two times: baseline (Ti) and one week after the 3rd bleaching session (Tf).

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene
* absence of active caries lesions
* never having undergone previous whitening therapy
* not present dental hypersensitivity
* don't be a smoker
* not be pregnant
* present at least 28 teeth in the oral cavity.

Exclusion Criteria:

* volunteers who were under orthodontic treatment,
* presence of periodontal disease
* dental cracks or fractures
* restorations and prostheses on anterior teeth
* extensive molar restorations
* gastroesophageal disorders
* severe internal dental darkening
* presence of dentinal exposure in anterior and / or posterior teeth.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Assessment of post bleaching sensitivity | 21 days
  For the assessment of postoperative sensitivity, patients were instructed to fill out a form to record tooth sensitivity daily, during the 21 days of treatment, based on individual pain perception. This form was delivered at each bleaching session, being returned to the researcher in the following session, that is, always one week after each bleaching session. The evaluation form consisted of the visual analogue scale (VAS). This scale consists of a 10 cm horizontal line, with scores of 0 and 10 at its ends, where 0 means no sensitivity and 10 means severe tooth sensitivity. The patient was instructed to draw a vertical line along the horizontal line of the scale, recording the intensity of tooth sensitivity per day. So that the distance in millimeters from the zero end could be later measured with the aid of a millimeter ruler, thus obtaining the patient's level of pain intensity.

SECONDARY OUTCOMES:
Color evaluation | Baseline (Ti) and one week after the 3rd whitening session (Tf).
  The VITA Easyshade spectrophotometer (VITA Zahnfabrik, Bad Säckingen, Germany) was used to measure the color, where the area of dental correspondence to be evaluated was the middle third of the buccal surface of the upper canines. To standardize the color readings, silicone trays were made, where the impression was extended from canine to canine. A window was created on the buccal surface of each canine of the silicone guide using a metal device with a 6 mm radius, corresponding to the diameter of the spectrophotometer tip. Thus, the tip of the device was inserted into the silicone guide to obtain the color parameters. Subsequently, the color difference between baseline (T i ) and one week after the 3rd bleaching session (T f ) was calculated using the CIEDE2000 formulas (ΔE00).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Para, Belém, Pará, Brazil